CLINICAL TRIAL: NCT06486103
Title: A Preliminary Investigation of the Safety and Effectiveness of Oral Probiotics Supplementation for Enhancing Vaginal Health in Females with Mild to Moderate Bacterial Vaginosis: an Open-Label, Single-Arm, Prospective Interventional Proof-of-Science Study.
Brief Title: A Clinical Study to Determine the Safety and Efficacy of an Oral Probiotic Supplementation to Improve Bacterial Vaginosis in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Meteoric Biopharmaceuticals Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator- Medical Director, NovoBliss Research Pvt Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB240018-MB
Record Dates: First submitted 2024-06-07; First posted 2024-07-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: An Open-Label, Single-Arm, Prospective Interventional Proof-of-Science Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bacterial Vaginosis (Experimental): Take one slow-release capsule twice a day, after meal, orally.
  Interventions: Other: MetSheFlora - Vaginal Health

INTERVENTIONS:
Other: MetSheFlora - Vaginal Health — Take one slow-release capsule twice a day, after meal.

SUMMARY:
A Preliminary Investigation of the Safety and Effectiveness of Oral Probiotics Supplementation for Enhancing Vaginal Health in Females with Mild to Moderate Bacterial Vaginosis: An Open-Label, Single-Arm, Prospective Interventional Proof-of-Science Study.

Total 14 healthy female patients aged 18 to 55 years with mild to moderate bacterial vaginosis will be enrolled to ensure 12 subjects complete the study.

DETAILED DESCRIPTION:
Potential subjects will undergo screening based on predefined inclusion and exclusion criteria only after obtaining written informed consent. The subject recruitment department will contact the potential subjects via telephone before the enrolment visit to confirm their participation.

Subjects shall be instructed to visit the facility for the following scheduled visits:

* Visit 01 [Day 01]: Screening, baseline evaluations, enrolment and test treatment dispensing.
* Visit 02 [Day 15 (±2 days)]: Treatment Phase, Follow-up Evaluations.
* Visit 03 [Day 30 (±2 days)]: Treatment End, Final Evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a healthy non-pregnant/non-lactating females aged 18 to 55 years.
2. Subjects having refrigerator at their home for storage of test treatment.
3. Presence of bacterial vaginosis (BV) as determined by gynaecological examination, including assessment for clinical symptoms such as abnormal vaginal discharge, malodour (moderate to very intense), and other relevant clinical indicators.
4. The subject is willing to provide written informed consent and follow study procedures.
5. The subject is willing to abide by the study protocol and restrictions, including abstaining from using any other intimate wash, lubricant, or treats during the study.
6. The subject is willing to use a highly effective method of contraception throughout the clinical investigation. This includes:

   1. Females of childbearing potential must practice and maintain an established method of birth control (e.g., IUD, diaphragm, condoms with spermicide, partner vasectomy, or abstinence).
   2. Non-childbearing potential females who are surgically sterile, post-menopausal for at least 1 year, or have had a tubal ligation, and agree to continue using the same contraception for the study duration.
7. Agreement for gynaecological pelvic examination by a Gynaecologist.
8. The subject is willing to abstain from sexual intercourse for a period of 24 hours before scheduled study visits to minimize potential interference with study assessments and measurements.

Exclusion Criteria:

1. The subject has used hormone replacement therapy in the last 3 months.
2. The subject has a history or visible evidence of chronic skin disease or regional infections, genital herpes, vaginal infections, or urinary tract infections.
3. The subject is pregnant/lactating, or are likely to become pregnant.
4. The subject has been diagnosed with or reported gynaecologic abnormalities within 60 days prior to study initiation that may influence study results.
5. The subject has severe systemic complications of viral infections, cardiovascular disorders, neurological disorders, renal disorders, or autoimmune disorders.
6. The subject has chronic infection/allergy/disease that may influence study results.
7. The subject has participated in clinical studies or received any investigational agent in the previous 30 days.
8. The subject has failed to satisfy the Investigator for fitness to participate for any other reason.
9. The subject has not experienced previous episodes of vaginal bleeding of unknown origin within the last 6 months of the screening visit.
10. The subject does not have vaginal prolapse and/or other medical conditions interfering with study conduct and participation.
11. The subject has not used systemic and/or local hormonal products for vaginal dryness or any other vaginal condition in the 3 months prior to screening

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy female patients aged 18 to 55 years with mild to moderate bacterial vaginosis.
Enrollment: 14 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Change in quality of vaginal discharge | On Day 01 (before administration) for baseline, and post-dose on Day 15 (±2 days) and Day 30 (±2 days)
  Assessment of the effectiveness of test treatment in terms of change in quality of vaginal discharge using 5 point scoring scale where 0 indicate absent and 4 indicates very intense
change in odour of vaginal discharge. | On Day 01 (before administration) for baseline, and post-dose on Day 15 (±2 days) and Day 30 (±2 days)
  Assessment of the effectiveness of test treatment in terms of change in odour of vaginal discharge using 5 point scoring scale where 0 indicate absent and 4 indicates very intense.
Nugent score | On Day 01 (before administration) for baseline, and post-dose on Day 30 (±2 days).
  Assessment of the effectiveness of test treatment in terms of change in Nugent score where 0-3 indicates normal, 4-6 indicates intermediate bacterial count and 7-10 indicates bacterial vaginosis.

SECONDARY OUTCOMES:
Change in vaginal pH | On Day 01 (before administration) for baseline, and post-dose on Day 15 (±2 days) and Day 30 (±2 days),
  Assessment of the effectiveness of test treatment in terms of change in vaginal pH
Change in VAS score | On Day 01 (before application) for baseline, and post-dose on Day 15 (±2 days) and Day 30 (±2 days).
  Assessment of the effectiveness of test treatment in terms of change in VAS score for vaginal itching where 0= indicates no itch and 10 indicates severe itch
Subject's perception | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of the subject's perception regarding the test treatment using a hedonic scale questionnaire for parameters such as smell, taste, overall palatability, perceived effectiveness.
Treatment-emergent adverse events (burning). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as burning.
Treatment-emergent adverse events (stinging). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as stinging using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (moisture). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as moisture using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (flaking). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as flaking using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (epithelial mucosa). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as epithelial mucosa using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (redness). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as redness using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (dryness). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as dryness.
Treatment-emergent adverse events (odour). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as odour using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (itching). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as itching using scoring scale 0= Indicate absent and 3= severe
Treatment-emergent adverse events (soreness of vulva ). | On Day 15 (±2 days) and Day 30 (±2 days) post-dose.
  Assessment of safety of test treatment through treatment-emergent adverse events such as soreness of vulva using scoring scale 0= Indicate absent and 3= severe
Safety laboratory tests including Haemoglobin | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Haemoglobin
Safety laboratory tests including Haematocrit | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Haematocrit
Safety laboratory tests including RBC count | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including RBC count
Safety laboratory tests including packed cell volume | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including packed cell volume
Safety laboratory tests including RBC morphology | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including RBC morphology
Safety laboratory tests including mean corpuscular volume | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including mean corpuscular volume
Safety laboratory tests including mean corpuscular hemoglobin | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including mean corpuscular hemoglobin
Safety laboratory tests including mean corpuscular haemoglobin concentration | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including mean corpuscular haemoglobin concentration
Safety laboratory tests including Red blood cell distribution width | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Red blood cell distribution width
Safety laboratory tests including Neutrophils | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Neutrophils
Safety laboratory tests including CBC (Lymphocytes) | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Lymphocytes
Safety laboratory tests including Eosinophils | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Eosinophils
Safety laboratory tests including Monocyte | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Monocyte
Safety laboratory tests including Basophils | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Basophils
Safety laboratory tests including Platelet count | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Platelet count
Safety laboratory tests including mean platelet volume | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including mean platelet volume
Safety laboratory tests including plateletcrit | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including plateletcrit
Safety laboratory tests including Platelet Distribution Width | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Platelet Distribution Width
Safety laboratory tests including random blood sugar | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including random blood sugar
Safety laboratory tests including Total serum cholesterol | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Total serum cholesterol
Safety laboratory tests including CBC (triglyceride) | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including triglyceride
Safety laboratory tests including high-density lipoprotein | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including high-density lipoprotein
Safety laboratory tests including low-density lipoprotein | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including low-density lipoprotein
Safety laboratory tests including CBC (Serum Creatinine) | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Serum Creatinine
Safety laboratory tests including Urinalysis | On Day 01 before dosing, and on Day 30 (±2 days) post-dose
  Assessment of safety of test treatment through the performance of safety laboratory tests including Urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No